CLINICAL TRIAL: NCT00123708
Title: Hypertonia in Patients With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050204; 05-CH-0204
Record Dates: First submitted 2005-07-23; First posted 2005-07-25 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-11-13

CONDITIONS: Cerebral Palsy; Muscle Hypertonia
Keywords: Spasticity; Dystonia; Movement Disorders; Walking; Muscle Weakness; Resistance; Gait; Cerebral Palsy; CP
MeSH Terms: conditions — Cerebral Palsy; Muscle Hypertonia; Muscle Spasticity; Dystonia; Movement Disorders; Muscle Weakness

SUMMARY:
This study will classify types of hypertonia in patients with cerebral palsy and determine if the classifications are reasonable in relation to the functional task of walking. Hypertonia is an abnormal increase in muscle tension. It is a common symptom of cerebral palsy that can lead to loss of function and deformity. This study may help scientists improve evaluation criteria for hypertonia and, ultimately, treatment results.

Patients with cerebral palsy who are older than 6 years of age may be eligible for this study. Candidates are screened with a medical history and clinical evaluation.

Participants are asked to walk in the lab while cameras record their movement. During this test, subjects wear a t-shirt and shorts with their arms and legs wrapped with a soft, rubber-like material. A piece of firm material is attached to the rubber sleeves and small plastic reflective balls are attached to the firm material. Balls may also be attached to the skin, using an adhesive. With the balls in place, the subject walks several times while cameras record the positions of the balls. In addition, small metal electrodes attached to the skin with an adhesive measure the electrical activity in the muscles.

After the walking test is completed, subjects' leg muscle strength is measured with a special device while they perform three activities. First, they sit on a special chair with their leg and foot placed in an apparatus that measures their strength, then lie on their back, then on their stomach, and then stand on one foot holding a bar to balance during part of one activity. During the activities, their reflexes are tested, they are asked to move their legs, and their legs are moved for them.

DETAILED DESCRIPTION:
Cerebral palsy (CP) affects 0.25% of newborn babies in the U.S. alone each year. Hypertonia (increased joint resistance to externally imposed motion) is a common symptom that limits function in this patient population. It may originate in spasticity, dystonia or rigidity or may be a combination of all these factors. Surgical, rehabilitation and pharmacotherapeutic methods are used to improve functional outcome in patients with cerebral palsy. These treatments are not always effective, and the amount of improvement is difficult to predict. The choice of treatment is based on clinical tests that are not objective, especially in children, and they do not allow for differentiation between various causes of increased joint resistance. As a result, ineffective treatments are offered to patients with different types of movement disorders. The complex torque devices used in research facilities to quantify the resistance of a joint cannot be easily applied in clinical settings. In previous studies, a portable measurement method was developed based on a hand-held force transducer, which allowed for the quantification of biomechanical and bioelectrical characteristics of resistance of a knee joint at different velocities. Using this method, we found different types of hypertonia that had not been previously reported in patients with cerebral palsy. It is not clear to what degree hypertonia restricts an ability to execute selected functional tasks, due in part to the considerable variability in patients with CP. If this variability could be decreased, the relationship between restricted ability and the different types of hypertonia would be easier to determine. Strong arguments exist to consider different pathophysiologies in these different types of hypertonia.

The aim of this non-invasive study is to sub-classify patients with CP based on the type of knee hypertonia, and to determine if the classification is valid during the functional tasks of walking. When validated, it can serve as a predictive model for the relationship between the clinical evaluation at bedside and functional outcome.

To classify hypertonia, the resistance of a knee joint at different velocities in knee flexion and extension and the maximum activation of stretched and shortened muscles are measured with a hand-held force transducer, an electrogoniometer, and surface electrodes in 100 patients with CP. The strength of velocity-dependent hypertonia during passive stretch and position, and/or velocity thresholds will be calculated. The knee extension and flexion muscles will be classified bilaterally as normal, or as one of the four types based on the pattern of activation of stretched muscles. To determine the impact of other impairments on the function, the maximum isometric knee flexion and extension strength and the monosynaptic reflexes of the rectus femoris muscle will be measured.

At the functional level, we will evaluate knee motion during walking. To determine the impact of hypertonia on function, the Spearman R correlation will be used to analyze data in patients within the same class. To determine if the classification holds during walking, the Cronbach's alpha coefficient will be calculated. The significance of differences will be tested at the level of significance alpha less than or equal to 0.05.

It is expected that as a result of this study, better criteria for classifying patients into predictable categories correlated to specific therapeutic responses will be established. In the future, the improvement of differential diagnoses with quantitative methods will increase the effectiveness of treatment by customizing the needs of each patient.

ELIGIBILITY:
* INCLUSION CRITERIA:

This study will include children and adult patients with cerebral palsy, patients with dystonia, and able-bodied children older than 6 years of age. Each patient must meet the following criteria:

The patient must have a diagnosis of cerebral palsy or dystonia

The patient must be able to follow the instructions to successfully complete the testing

The patient must be properly motivated and willing to do the tasks.

The patient must be older than 6 years

The patient must score a 2 or 3 on the walking subsection of the Gross Motor Function Classification System (GMFCS).

The patient must cease taking medications known to affect spasticity at least 48 hours before the first investigation; however, if any antispasticity medication is longstanding and stable it should be maintained during the entire study.

EXCLUSION CRITERIA:

Inability of the patient to follow the instructions to accomplish the task.

Structural deformities at the level of a knee joint.

If patients are unable to complete all the tasks or conditions they can still be enrolled to complete part of the study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2005-07-19; Primary Completion 2009-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] ASHWORTH B. PRELIMINARY TRIAL OF CARISOPRODOL IN MULTIPLE SCLEROSIS. Practitioner. 1964 Apr;192:540-2. No abstract available. PMID 14143329
- [Background] Barry MJ, VanSwearingen JM, Albright AL. Reliability and responsiveness of the Barry-Albright Dystonia Scale. Dev Med Child Neurol. 1999 Jun;41(6):404-11. doi: 10.1017/s0012162299000870. PMID 10400175
- [Background] Blackburn M, van Vliet P, Mockett SP. Reliability of measurements obtained with the modified Ashworth scale in the lower extremities of people with stroke. Phys Ther. 2002 Jan;82(1):25-34. doi: 10.1093/ptj/82.1.25. PMID 11784275